CLINICAL TRIAL: NCT05618197
Title: The Effects of Chronic Passive Heating on Vascular Function, Cognitive Function, Muscle Function and Heat Shock Protein Responses in Middle-aged to Older Adults: A Randomised, Controlled Crossover Trial
Brief Title: Chronic Passive Heating in Healthy Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Portsmouth (Other)
Responsible Party: Principal Investigator, Ant Shepherd, Senior Lecturer, University of Portsmouth
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: UoPCPHHOA
Record Dates: First submitted 2022-11-08; First posted 2022-11-16 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-03

CONDITIONS: Aging
Keywords: Passive heating; Endothelial function; Heat shock proteins; Cognitive function; Muscle strength

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Passive heating intervention (Experimental): ~3x per week of 1 h hot water immersion (to the clavicle, @40°C, rectal temperature ~38.5°C and <39°C) sessions over a period of 6 weeks.
  Interventions: Other: Passive heating
- Control (No Intervention): 6 weeks of no hot water immersion

INTERVENTIONS:
Other: Passive heating — ~3x per week of 1 h hot water immersion (to the clavicle, @40°C, rectal temperature ~38.5°C and <39°C) sessions over a period of 6 weeks.
  Arms: Passive heating intervention

SUMMARY:
Aging is associated with a decline in cardiovascular health, cognitive function and losses in muscle strength, with half or more of those over age 65 suffering from two or more comorbidities (e.g., heart disease, type 2 diabetes). The worldwide population of older adults is growing rapidly, with one in six people expected to be over age 65 by 2050. This will place further financial burden from chronic diseases on already stressed healthcare systems. While studies show that frequent exercise is an effective way for older adults to maintain or improve cardiovascular and metabolic health, older individuals are less physically active and do not adhere well to exercise programs, often due to physical or medical limitations. Therefore, alternative methods for older adults to get the same health benefits as exercise require further exploration. Recent work has shown that passive heat therapy may be one such alternative solution.

DETAILED DESCRIPTION:
Aging is associated with declines in cardiovascular health and cognitive function as well as chronic inflammation and the development of neurodegenerative conditions such as Alzheimer's and Parkinson's disease. Additionally, ageing results in a loss of muscle size and strength, commonly referred to as sarcopenia, leading to increased risk of falls or adverse exercise-related events. It is well understood that frequent exercise improves cardiovascular and metabolic health whilst lowering the risk of disease and all-cause mortality, acting as a treatment for many different health conditions. Despite the evidence of its efficacy, many individuals struggle with adherence to exercise programmes, particularly older adults and clinical populations, with many individuals within these populations unable to perform exercise due to physical limitations or medical contraindications. With one in six people expected to be over the age of 65 years by 2050 and corresponding increases in non-communicable diseases (e.g., cancer, diabetes, cardiovascular disease) anticipated from this aging population, the development of adjunct treatments or alternatives to exercise to improve general health in older populations is needed.

Recent work has shown that a potential solution could be the use of passive heat therapy (PHT) (e.g., hot water immersion, sauna), which can achieve health benefits comparable to exercise. Previous work by Brunt and colleagues using eight weeks of chronic heat therapy has demonstrated systemic macro- and microvascular adaptations in young, healthy individuals including improved endothelial function, reduced arterial stiffness and cutaneous vascular conductance. Chronic passive heat acclimation in young, healthy adults has also been shown to improve working memory. Additional studies have shown that ten weeks of passive heating improved muscle strength in middle-aged men and ten days of daily pulsed shortwave diathermy attenuated immobilization-induced muscle atrophy in young, healthy adults.

One potential mechanism for the physiological benefits obtained from PHT is the increase of cytoprotective heat shock proteins (HSP) (specifically HSP27, HSP60, HSP70 and HSP90) intracellularly (i) and extracellularly (e) in response to increases in deep body temperature. Increases in the expression of these HSPs have been shown to play a role in reducing inflammation and protecting the vasculature via increases in endothelial nitric oxide synthase activity. Increased HSP concentrations may also prevent the accumulation of harmful biomarkers in the brain that play a role in cognitive decline and development of neurodegenerative diseases. Aging, however, is associated with a reduction in HSP transcription activity in various tissues, resulting in an impaired heat shock response and development of a pro-inflammatory state. Previous work using acute hot water immersion has shown increases in eHSP70. The only study to test the effects of chronic hot water immersion on resting iHSP70 showed no effect, however, the magnitude of stimulus (39°C water) applied by Hoekstra and colleagues and the resultant changes in core temperature were likely too low to induce any changes in HSPs.

These studies provide promising evidence that health benefits from PHT similar to those from exercise could translate to older adults. However, most studies testing the effects of PHT on humans have been performed in young, healthy adults, whereas older individuals are likely to derive the greatest benefit from any positive effects of PHT. To date, no study has examined the longer-term effects of PHT on macrovascular, microvascular, cognitive or muscle function, or HSPs in older adults. Therefore, further research is needed to confirm that heat therapy confers the same beneficial health adaptations in older adults.

ELIGIBILITY:
Inclusion Criteria:

* Male or female age ≥ 55
* Free from cardiometabolic disease
* Body mass index of 18-35 kg/m2
* Receipt of a normal 12-lead ECG approved by the School Independent Medical Officer
* Capacity to understand and provide their written, informed consent to participate in the study protocol

Exclusion Criteria:

* Unable to understand or cooperate with the study protocol due to learning difficulties or otherwise
* Any current, or past medical (last five years), history of any cardiovascular, respiratory, cancer, renal, hepatic, gastrointestinal, haematological, lymphatic, neurological, psychiatric, or any other disease or diseases.
* Any regular medication for the last five years (not including acute courses of treatment of less than one month for discrete, resolved conditions).
* Medications that may influence physiological responses to the passive heating intervention Uncontrolled hypertension (≥ 150 mmHg systolic and/or ≥ 90 mmHg diastolic)
* Body mass index of > 35 kg/m2
* Recent long-term exposure to a hot climate (within the previous three months)
* Current smoker (or have stopped smoking within the previous three months)

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2023-05-23 (Actual); Primary Completion 2025-06-06 (Actual); Study Completion 2025-06-06 (Actual)

PRIMARY OUTCOMES:
Brachial artery flow-mediated dilation | Pre and post 6 weeks of passive heating and pre and post 6 weeks no intervention with 6 weeks washout between arms
  Percentage change from baseline in brachial artery diameter assessed by ultrasound.

SECONDARY OUTCOMES:
Brachial and carotid artery blood flow velocity | Pre and post 6 weeks of passive heating and pre and post 6 weeks no intervention with 6 weeks washout between arms
  Change from baseline in blood flow velocity of the brachial artery and right common carotid artery as assessed via ultrasound. cm/s is the unit.
Carotid vessel diameter | Pre and post 6 weeks of passive heating and pre and post 6 weeks no intervention with 6 weeks washout between arms
  Change from baseline in vessel diameter of the right common carotid artery as assessed via ultrasound. mm is the unit.
Carotid intima-media thickness | Pre and post 6 weeks of passive heating and pre and post 6 weeks no intervention with 6 weeks washout between arms
  Change from baseline in intima-media thickness of the right common carotid artery as assessed via ultrasound. mm is the unit
Carotid compliance | Pre and post 6 weeks of passive heating and pre and post 6 weeks no intervention with 6 weeks washout between arms
  Change in compliance of the right common carotid artery and return to baseline as assessed via ultrasound. µm^2 per kilopascal is the unit.
Carotid distensibility | Pre and post 6 weeks of passive heating and pre and post 6 weeks no intervention with 6 weeks washout between arms
  Change in distensibility of the right common carotid artery and return to baseline as assessed via ultrasound. 10^-3/kPa is the unit.
Carotid stiffness | Pre and post 6 weeks of passive heating and pre and post 6 weeks no intervention with 6 weeks washout between arms
  Change in stiffness of the right common carotid artery and return to baseline as assessed via ultrasound. Meters per second is the unit.
Microvascular function | Pre and post 6 weeks of passive heating and pre and post 6 weeks no intervention with 6 weeks washout between arms
  Change from baseline in microvascular function as assessed via iontophoresis on the forearm with acetylcholine (ACh) and Insulin, Area under the curve is the unit.
Stroke volume | Pre and post 6 weeks of passive heating and pre and post 6 weeks no intervention with 6 weeks washout between arms
  Change from baseline in stroke volume measured noninvasively via thoracic impedance. mL/m^2 is the unit
Total peripheral resistance | Pre and post 6 weeks of passive heating and pre and post 6 weeks no intervention with 6 weeks washout between arms
  Change from baseline in total peripheral resistance measured noninvasively via thoracic impedance.
Cardiac output | Pre and post 6 weeks of passive heating and pre and post 6 weeks no intervention with 6 weeks washout between arms
  Change from baseline in cardiac output measured noninvasively via thoracic impedance. L/min is the unit.
Mean arterial pressure | Pre and post 6 weeks of passive heating and pre and post 6 weeks no intervention with 6 weeks washout between arms
  Change from baseline in resting mean arterial pressure. mmHg is the unit.
Systolic blood pressure | Pre and post 6 weeks of passive heating and pre and post 6 weeks no intervention with 6 weeks washout between arms
  Change from baseline in resting systolic blood pressure. mmHg is the unit.
Diastolic blood pressure | Pre and post 6 weeks of passive heating and pre and post 6 weeks no intervention with 6 weeks washout between arms
  Change from baseline in resting diastolic blood pressure. mmHg is the unit.
Intracellular HSP27 concentration | Pre and post 6 weeks of passive heating and pre and post 6 weeks no intervention with 6 weeks washout between arms
  Change from baseline in resting iHSP27 concentrations? Measured via immunoblotting in peripheral blood mononuclear cells (PBMCs).
Intracellular HSP60 concentration | Pre and post 6 weeks of passive heating and pre and post 6 weeks no intervention with 6 weeks washout between arms
  Change from baseline in resting iHSP60 concentrations? Measured via immunoblotting in peripheral blood mononuclear cells (PBMCs).
Intracellular HSP70 concentration | Pre and post 6 weeks of passive heating and pre and post 6 weeks no intervention with 6 weeks washout between arms
  Change from baseline in resting iHSP70 concentrations? Measured via immunoblotting in peripheral blood mononuclear cells (PBMCs).
Intracellular HSP90 concentration | Pre and post 6 weeks of passive heating and pre and post 6 weeks no intervention with 6 weeks washout between arms
  Change from baseline in resting iHSP90 concentrations? Measured via immunoblotting in peripheral blood mononuclear cells (PBMCs).
Plasma eHSP27 concentration | Pre and post 6 weeks of passive heating and pre and post 6 weeks no intervention with 6 weeks washout between arms
  Change from baseline in resting plasma eHSP27 concentrations? Measured via ELISA
Plasma eHSP60 concentration | Pre and post 6 weeks of passive heating and pre and post 6 weeks no intervention with 6 weeks washout between arms
  Change from baseline in resting plasma eHSP60 concentrations? Measured via ELISA.
Plasma eHSP70 concentration | Pre and post 6 weeks of passive heating and pre and post 6 weeks no intervention with 6 weeks washout between arms
  Change from baseline in resting plasma eHSP70 concentrations? Measured via ELISA.
Plasma eHSP90 concentration | Pre and post 6 weeks of passive heating and pre and post 6 weeks no intervention with 6 weeks washout between arms
  Change from baseline in resting plasma eHSP90 concentrations? Measured via ELISA.
Reaction time | Pre and post 6 weeks of the passive heating intervention during the first and final heating visits at time points of pre-hot water immersion, 0 hours post and 3 hours post hot water immersion
  Change in reaction time in response to a heating challenge. Assessed using ANAM: Automated Neurophysiological Assessment Metrics.
Logical reasoning | Pre and post 6 weeks of the passive heating intervention during the first and final heating visits at time points of pre-hot water immersion, 0 hours post and 3 hours post hot water immersion
  Change in logical reasoning in response to a heating challenge. Assessed using ANAM: Automated Neurophysiological Assessment Metrics.
Memory | Pre and post 6 weeks of the passive heating intervention during the first and final heating visits at time points of pre-hot water immersion, 0 hours post and 3 hours post hot water immersion
  Change in memory in response to a heating challenge. Assessed using ANAM: Automated Neurophysiological Assessment Metrics.
Cerebral oxygenation | Pre and post 6 weeks of the passive heating intervention during the first and final heating visits at time points of pre-hot water immersion, 0 hours post and 3 hours post hot water immersion
  Change in cerebral oxygenation in response to a heating challenge. Assessed using Near-infrared spectroscopy (NIRS) attached to the forehead.
Maximum quadriceps strength | Pre and post 6 weeks of passive heating and pre and post 6 weeks no intervention with 6 weeks washout between arms
  Change from baseline in quadriceps strength. Assessed using an isokinetic dynamometer.
Maximum grip strength | Pre and post 6 weeks of passive heating and pre and post 6 weeks no intervention with 6 weeks washout between arms
  Change from baseline in grip strength. Assessed using a hand grip dynamometer.
Lower extremity function | Pre and post 6 weeks of passive heating and pre and post 6 weeks no intervention with 6 weeks washout between arms
  Change from baseline in lower extremity function. Assessed using the Short Physical Performance Battery (balance, walking speed and sit to stand) .
Quadriceps muscle electrical activity | Pre and post 6 weeks of passive heating and pre and post 6 weeks no intervention with 6 weeks washout between arms
  Change from baseline in quadriceps muscle electrical activity. Assessed using electromyography (EMG) on the vastus lateralis of the dominant leg.
Balance capacity | Pre and post 6 weeks of passive heating and pre and post 6 weeks no intervention with 6 weeks washout between arms
  Does chronic passive heating improve balance? Assessed using motion capture and force plates.
Gait characteristics | Pre and post 6 weeks of passive heating and pre and post 6 weeks no intervention with 6 weeks washout between arms
  Change from baseline in gait characteristics. Assessed using motion capture and force plates.
Total minutes of physical activity (light, moderate, moderate to vigorous physical activity). | Pre and during the final week of 6 weeks of passive heating and pre and during the final week of 6 weeks no intervention with 6 weeks washout between arms
  Change from baseline in physical activity levels. Assessed using wrist-worn accelerometry.
Sleep efficiency (time in bed + time asleep) | Pre and during the final week of 6 weeks of passive heating and pre and during the final week of 6 weeks no intervention with 6 weeks washout between arms
  Change from baseline in sleep efficiency. Assessed using wrist-worn accelerometry.

CONTACTS AND LOCATIONS:
Overall Officials: Zoe Saynor, PhD, Study Director — University of Portsmouth
Locations (1):
- Spinnaker Building, Portsmouth, Hampshire, United Kingdom